CLINICAL TRIAL: NCT04977752
Title: Quality of Life in Patients With Hirschsprung's Disease in Relation to Surgical Technique: a Study of a Danish Population
Brief Title: Hirschsprung's Disease: Surgical Techniques and Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christoffer Cain Hansen, Student, University of Southern Denmark
Other Study IDs: 232-2021-NQ
Record Dates: First submitted 2021-07-21; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study examining the long-term quality of life in patients with Hirschsprung's Disease in relation to the choice of surgical technique.

DETAILED DESCRIPTION:
Hirschsprung's Disease (HD) is a developmental defect causing functional obstruction of bowel. It is a condition that almost always requires surgical intervention. This study aims to examine the relation between quality of life and surgical technique in patients with Hirschsprung's disease in hopes of providing insight into advantages and disadvantages of different surgical techniques employed at OUH, department for general surgery in the time between 1985 and 2012. This will be done based on answers given on a set of validated questionnaires that has been sent to all patients diagnosed with HD in the years 1985 to 2012 at OUH, department for general surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with HD at the Surgical Department at Odense University Hospital from 1985 to 2012 will be invited to enroll in the study.

Exclusion Criteria:

* lack of informed consent, pregnancy, wrong diagnosis and inability to understand or answer the questionnaires.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with HD at OUH, department for general surgery between 1985 and 2012.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-01-14 (Estimated); Study Completion 2022-01-14 (Estimated)

PRIMARY OUTCOMES:
Hirschsprung Quality of life Questionnaire sub scales and total score | Day 1
  Disease specific questionnaire including sub scales for laxative and constipating diet, presence of diarrhoea and constipation, faecal and urinary incontinence, social and emotional functioning, body image, physical symptoms and sexual functioning. Each item is phrased as a multiple-choice question with four response options; never, once in a while, often and very often. Responses are linearly transformed on a 0-100 scale with a higher score indicating better QOL.
General Quality of Life | Day 1
  Based on a generic SF-36 questionnaire subscaled into perception of health, physical functioning, physical role functioning, emotional functioning and emotional role functioning. Each question is phrased as a multiple-choice question with varying options depending on the type of question.
Type of Surgical Intervention | Day 1
  At our centre three different types of surgical approaches have been employed: Soave operation, Low anterior resection (Rehbeins operation) and trans-anal pullthrough. These outcomes will be correlated to outcomes of quality of life in other to compare the resulting quality of life between the different surgical approaches.

SECONDARY OUTCOMES:
Rate of Complications | Day 1
  Data will be retrieved through electronic medical journals. Data such as short term and long term major postoperative complications will be gathered in order to compare prevalence of surgical complications to type of surgical approach.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Fyn, Denmark